CLINICAL TRIAL: NCT07109505
Title: Comparison of Clinical and Patient Centered Outcomes: Postoperative Multi-nutrient Meal Plus Enhanced Recovery vs. Enhanced Recovery Alone
Brief Title: Nutrition to Support Postoperative Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Hitchcock Foundation (Other)
Responsible Party: Principal Investigator, Stacie.G.Deiner, LeRoy Garth Professor and Vice Chair for Research, Department of Anesthesiology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY02002743
Record Dates: First submitted 2025-06-25; First posted 2025-08-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Care; Postoperative Complications; Cognition; Nutritional Assessment; Nutritional Intervention
Keywords: Nutrition; Postoperative; Cognition
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: The randomization assignment will consist of two groups: Shake and instructions or instructions only.
Who Masked: Investigator
Masking Description: The randomization assignment (shake and instructions or instructions only) will not be double blinded since the participants will know if they receive a shake mix or not. However, the coordinator performing assessments after discharge will be blinded to group. A separate, unblinded study team member will track compliance (see above).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shake and instructions (Experimental): For the intervention arm, an unblinded study team member will deliver and review the Nutrition After Surgery and postoperative supplementation instructions with the participant.
  Additionally, an unblinded study team member will give each participant a 30-day supply of single-servings. They will be instructed to consume 1 packet per day for 30 days, reconstituted per instructions (see instructions file), after discharge from the hospital. The unblinded researchers will work with the coordinator team to provide participants with a plan for supplementation (normal or underweight participants) or meal replacement (overweight or obese patients). Participants will be instructed to keep track of their shake consumption on a daily basis. Shake consumption logs will be collected via REDCap surveys sent to participants and reviewed by the unblinded coordinators/investigators for adverse events and compliance.
  Interventions: Dietary Supplement: Nutritional Shake
- Nutrition Instructions Only (Other): The control arm receives the Nutrition After Surgery instructions, which provide guidelines for healthy eating after surgery but not the nutritional shake. The intervention arm receives the same instructions along with the nutrition shake mix and accompanying postoperative supplementation
  Interventions: Other: Nutritional Instructions Only

INTERVENTIONS:
Dietary Supplement: Nutritional Shake — The shake mixes will be dry shelf -stable powders prepared with ingredients readily available in the US food supply and contain a minimum of 990 mg total cocoa flavanols, with a profile to support general nutritional health including 10 g protein. Accordingly, each shake contains approximately 95 mg of caffeine, equivalent to a medium-sized cup of coffee. Based on prior studies of cognition, additional composition specifications are: 1600 mg DHA and up to 400 mg EPA and 550 mg choline; >250 mg epicatechin and epigallocatechin (plant polyphenols); multivitamin/mineral fortification to ensure 50-100% of all essential micronutrients except calcium (to prevent competitive absorption with other divalent cations). Participants will be given a supply of pre-portioned daily servings upon discharge from the hospital, for 30 days after surgery.
  Arms: Shake and instructions
Other: Nutritional Instructions Only — The control arm receives the Nutrition After Surgery instructions, which provide guidelines for healthy eating after surgery but not the nutritional shake. The intervention arm receives the same instructions along with the nutrition shake mix and accompanying postoperative supplementation
  Arms: Nutrition Instructions Only

SUMMARY:
Older surgical patients commonly have malnutrition, and there is evidence these patients have increased risk for poor physical and brain recovery after surgery and anesthesia. There are scientific-based recommendations to provide nutritional supplements to support recovery. However, to date these recommendations do not address a broad group of nutrients likely to reverse common deficiencies. Team members have created a palatable, broad-spectrum and stable nutritional shake that we will give to patients after surgery. We propose to test the nutritional shake in frail older surgical patients at Dartmouth Health to determine if a nutrition shake provided after surgery improves recovery of physical function and cognitive abilities. Half the patients will receive the shake and the other will receive the standard of care postoperative nutritional instructions after surgery. We will collect information regarding physical function and cognitive abilities of all the patients while in the hospital and 90 days after surgery. We will use this data to apply for funding for a powered randomized trial to determine the role of nutrition in optimizing physical and cognitive recovery from surgery in older patients.

DETAILED DESCRIPTION:
We will recruit a cohort of community dwelling patients, age 70 years and older for elective major abdominal and orthopedic surgery. Demographics, medical history, medications will be obtained from the electronic health record and confirmed with the patient. Patients randomized to the nutrition shake arm will receive a provided daily nutritional shake (starting when they leave the hospital and for 1-month after hospital discharge). The shake consists of a comprehensive panel of essential nutrients to support maintenance of muscle, metabolic and brain health.

ELIGIBILITY:
Inclusion Criteria:

* patients >=70 years old having major orthopedic or abdominal surgery, defined as a procedure with a planned inpatient stay of at least one night.

Exclusion Criteria:

* emergency surgery, diagnosis of dementia or major psychiatric diagnosis such as schizophrenia, Parkinson's disease, inability to consent for themselves, unwilling or unable to complete all study requirements and measurements, any known food allergy, dislike of shake flavor(s), unwilling or unable to tolerate caffeine in shake, unable to take oral nutrition, BMI >45, diagnosis of an eating disorder, insulin dependent diabetes.
* MRI procedure eligibility will be assessed using the DHMC Department of Radiology's standard MRI Safety Checklist, which screens for potential contraindications to MRI scanning such as metal in the body, possible exposure to metal in the eyes, pregnancy, and claustrophobia. Any individual with a contraindication to MRI scanning will not be eligible to participate in the optional MRI component.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Aim 1a: Postoperative change in disability scores | 90 days
  This aim will compare postoperative change in disability scores, as measured by World Health Organization Assessment Schedule 2.0 (WHODAS 2.0), from baseline to 1 month and baseline to 3 months. Results will be scored on a 5-point Likert scale and summed to a total score ranging 0 to 100, where 0 indicates no disability and 100 indicates full disability. The outcome will compare patients receiving a 30-day supply of daily nutritional shake and general healthy nutrition recommendations versus those only receiving general healthy nutrition recommendations without a provided shake
Aim 1b: Postoperative change in cognitive function | 90 days
  This aim will compare postoperative change in cognitive function, as measured by The Montreal Cognitive Assessment (T-MoCA), from baseline to 1 month and baseline to 3 months. Scores will range from 0 to 30 points, with higher scores indicating greater cognitive function. The outcome will compare patients receiving a 30-day supply of a daily nutritional shake and general healthy nutritional recommendations versus those receiving only healthy nutritional recommendations without a provided shake.

OTHER OUTCOMES:
Banking of blood specimens for future analysis | day of surgery and postoperative day 1
  Mechanistic investigations of effects of multi-component nutrition food (MCN). We will collect and freeze blood specimens for a secondary analysis of blood markers of neural injury and inflammation that has been observed in surgical cohorts. No analysis of the samples will be performed currently. We will measure the proportion of patients with samples on the day of surgery and at postoperative day one.
Feasibility of MRI scan 30 days after surgery | 30 days after surgery
  As part of the pilot, we will obtain imaging on a small subset of participants, working together with the DH Department of Psychiatry Brain Imaging Lab, to allow us pursue a mechanistic line of inquiry in future applications. The measure of success is the proportion of patients eligible and willing vs. the number approached, and the proportion of patients who consent to the MRI who successfully complete the hour- long protocol. We will ask patients about whether they are willing to participate in the postoperative MRI until we have 4 patients who are eligible and willing to complete the imaging protocol, which will include anatomical MRI, resting state and task based functional MRI, diffusion tensor imaging, and arterial spin labeling.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie G Deiner, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
The consent does not ask participants to share their data outside the study

REFERENCES:
- [Background] Katz MJ, Wang C, Nester CO, Derby CA, Zimmerman ME, Lipton RB, Sliwinski MJ, Rabin LA. T-MoCA: A valid phone screen for cognitive impairment in diverse community samples. Alzheimers Dement (Amst). 2021 Feb 5;13(1):e12144. doi: 10.1002/dad2.12144. eCollection 2021. PMID 33598528
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Katz S. Assessing self-maintenance: activities of daily living, mobility, and instrumental activities of daily living. J Am Geriatr Soc. 1983 Dec;31(12):721-7. doi: 10.1111/j.1532-5415.1983.tb03391.x. PMID 6418786
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Mendoza TR, Chen C, Brugger A, Hubbard R, Snabes M, Palmer SN, Zhang Q, Cleeland CS. The utility and validity of the modified brief pain inventory in a multiple-dose postoperative analgesic trial. Clin J Pain. 2004 Sep-Oct;20(5):357-62. doi: 10.1097/00002508-200409000-00011. PMID 15322443
- [Background] Pavlin DJ, Sullivan MJ, Freund PR, Roesen K. Catastrophizing: a risk factor for postsurgical pain. Clin J Pain. 2005 Jan-Feb;21(1):83-90. doi: 10.1097/00002508-200501000-00010. PMID 15599135
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Berger MM, Amrein K, Barazzoni R, Bindels L, Breton I, Calder PC, Cappa S, Cuerda C, D'Amelio P, de Man A, Delzenne NM, Forbes A, Genton L, Gombart AF, Joly F, Laviano A, Matthys C, Phyo PP, Ravasco P, Serlie MJ, Shenkin A, Stoffel NU, Talwar D, van Zanten ARH. The science of micronutrients in clinical practice - Report on the ESPEN symposium. Clin Nutr. 2024 Jan;43(1):268-283. doi: 10.1016/j.clnu.2023.12.006. Epub 2023 Dec 9. PMID 38104489
- [Background] Norman K, Hass U, Pirlich M. Malnutrition in Older Adults-Recent Advances and Remaining Challenges. Nutrients. 2021 Aug 12;13(8):2764. doi: 10.3390/nu13082764. PMID 34444924
- [Background] Valletta M, Vetrano DL, Calderon-Larranaga A, Kalpouzos G, Canevelli M, Marengoni A, Laukka EJ, Grande G. Association of mild and complex multimorbidity with structural brain changes in older adults: A population-based study. Alzheimers Dement. 2024 Mar;20(3):1958-1965. doi: 10.1002/alz.13614. Epub 2024 Jan 3. PMID 38170758
- [Background] Roberts SB, Franceschini MA, Silver RE, Taylor SF, de Sa AB, Co R, Sonco A, Krauss A, Taetzsch A, Webb P, Das SK, Chen CY, Rogers BL, Saltzman E, Lin PY, Schlossman N, Pruzensky W, Bale C, Chui KKH, Muentener P. Effects of food supplementation on cognitive function, cerebral blood flow, and nutritional status in young children at risk of undernutrition: randomized controlled trial. BMJ. 2020 Jul 22;370:m2397. doi: 10.1136/bmj.m2397. PMID 32699176
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Williams DGA, Villalta E, Aronson S, Murray S, Blitz J, Kosmos V, Wischmeyer PE; Duke Perioperative Enhancement Team (POET). Tutorial: Development and Implementation of a Multidisciplinary Preoperative Nutrition Optimization Clinic. JPEN J Parenter Enteral Nutr. 2020 Sep;44(7):1185-1196. doi: 10.1002/jpen.1824. Epub 2020 Mar 31. PMID 32232882
- [Background] Williams JD, Wischmeyer PE. Assessment of perioperative nutrition practices and attitudes-A national survey of colorectal and GI surgical oncology programs. Am J Surg. 2017 Jun;213(6):1010-1018. doi: 10.1016/j.amjsurg.2016.10.008. Epub 2016 Nov 17. PMID 27889271
- [Background] Fried TR, Tinetti ME, Iannone L, O'Leary JR, Towle V, Van Ness PH. Health outcome prioritization as a tool for decision making among older persons with multiple chronic conditions. Arch Intern Med. 2011 Nov 14;171(20):1854-6. doi: 10.1001/archinternmed.2011.424. Epub 2011 Sep 26. No abstract available. PMID 21949032
- [Background] Becher RD, Vander Wyk B, Leo-Summers L, Desai MM, Gill TM. The Incidence and Cumulative Risk of Major Surgery in Older Persons in the United States. Ann Surg. 2023 Jan 1;277(1):87-92. doi: 10.1097/SLA.0000000000005077. Epub 2021 Jul 14. PMID 34261884
- [Background] Deiner S, Baxter MG, Mincer JS, Sano M, Hall J, Mohammed I, O'Bryant S, Zetterberg H, Blennow K, Eckenhoff R. Human plasma biomarker responses to inhalational general anaesthesia without surgery. Br J Anaesth. 2020 Sep;125(3):282-290. doi: 10.1016/j.bja.2020.04.085. Epub 2020 Jun 11. PMID 32536445
- [Background] Evered L, Silbert B, Scott DA, Zetterberg H, Blennow K. Association of Changes in Plasma Neurofilament Light and Tau Levels With Anesthesia and Surgery: Results From the CAPACITY and ARCADIAN Studies. JAMA Neurol. 2018 May 1;75(5):542-547. doi: 10.1001/jamaneurol.2017.4913. PMID 29459944